CLINICAL TRIAL: NCT00879398
Title: Post Marketing Surveillance Study To Observe Safety And Efficacy Of Toviaz (Registered)
Brief Title: Toviaz Post Marketing Surveillance Study
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A0221075
Record Dates: First submitted 2009-04-09; First posted 2009-04-10 (Estimated); Results first posted 2015-09-04 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-09

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- OAB-Toviaz: All patients who enrolled in this study
  Interventions: Drug: Toviaz treatment

INTERVENTIONS:
Drug: Toviaz treatment — 4 mg starting then can be followed by 8 mg

SUMMARY:
The objective of this study is to determine the problems and questions of safety and efficacy of Toviaz® under the standard conditions of usage.

DETAILED DESCRIPTION:
continuous registration method

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are diagnosed as Overactive Bladder (OAB) defined as urgency, with or without urgency incontinence, usually with frequency and nocturia, in the absence of local or metabolic factors explaining these factors.

Exclusion Criteria:

* Hypersensitivity to the active substance or to peanut or soya or any of the excipients
* Urinary retention
* Gastric retention
* Uncontrolled narrow angle glaucoma
* Myasthenia gravis
* Severe hepatic impairment (Child Pugh C)
* Concomitant use of potent CYP3A4 inhibitors in subjects with moderate to severe hepatic or renal impairment
* Severe ulcerative colitis
* Toxic megacolon
* Patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption (Toviaz® prolonged-release tablets contain lactose)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Subjects who are diagnosed as Overactive Bladder (OAB) defined as urgency, with or without urgency incontinence, usually with frequency and nocturia, in the absence of local or metabolic factors explaining these factors.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2009-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (79):
- South Korea (79):
  - Soo Urology Clinic, Asan, Chungcheongnam-do
  - Seo Kyung-Keun Urology Clinic, Cheonan-si, Chungcheongnam-do
  - Cheonan Medical Center, Cheonan-Si, Chungcheongnam-do
  - Seoul Urology Clinic, Gongju, Chungcheongnam-do
  - Lee Urology Clinic, Gongju, Chungcheongnam-do
  - Moa gynecology, Nonsan, Chungcheongnam-do
  - Song In-Ho Urology Clinic, Tangjin, Chungcheongnam-do
  - Jung Woong Gyo Urology Clinic, Wŏnju, Gangwon-do
  - Ansan Themapark Medical Center, Ansan, Gyeonggi-do
  - Woosung Yusung Hospital, Ansan, Gyeonggi-do
  - Kim Tae Joon Internal Medicine, Ansan-si, Gyeonggi-do
  - Yoo And Lee Dematology Urology Clinic, Bucheon-si, Gyeonggi-do
  - Myung Urology Hospital, Bucheon-si, Gyeonggi-do
  - Gimpo Woori Hospital, Gimpsi, Gyeonggi-do
  - Samsung Clinic, Goyang-si, Gyeonggi-do
  - Hwang Family Medicine Clinic, Goyang-si, Gyeonggi-do
  - Lee Urology Clinic, Namyangju, Gyeonggi-do
  - Park Dermatology And Urology Clinic, Pyeongtaek-si, Gyeonggi-do
  - Good morning Clinic, Pyeongtaek, Pyeongtaek-si, Gyeonggi-do
  - Cheong Urology Clinic, Seongnam-si, Gyeonggi-do
  - Na Seung Soo Urology Clinic, Seongnam-si, Gyeonggi-do
  - Good Urology Clinic, Seongnam-si, Gyeonggi-do
  - Seoul Urology Clinic, Seongnam-si, Gyeonggi-do
  - Bes Top Urology Clinic, Seongnam-si, Gyeonggi-do
  - Dongsuwon General Hospital, Suwon, Gyeonggi-do
  - Kim Dae Sung Clinic, Uijeongbu-si, Gyeonggi-do
  - Johan Urology Clinic, Uijeongbu-si, Gyeonggi-do
  - Min Urology Clinic, Uijeongbu-si, Gyeonggi-do
  - Choi Won Suk urology clinic, Yongin-si, Gyeonggi-do
  - Haram Urology Clinic, Yongin-si, Gyeonggi-do
  - Well Urology Clinic, Yongin, Gyeonggi-do
  - Hankook General Hospital, Cheongju-si, North Chungcheong
  - Shin Urology Clinic, Cheongju-si, North Chungcheong
  - Lee Urology Clinic, Yeongdong-gun, North Chungcheong
  - Chung Duck Young Urology Clinic, Daejeon
  - Yeonhap Urology Clinic, Daejeon
  - Taepyung urology clinic, Daejeon
  - Ssen Urology Clinic, Daejeon
  - Kim Se Gyeom Urology Clinic, Daejeon
  - Kwon Urology Clinic, Daejeon
  - Incheon Medical Center, Incheon
  - Incheonsarang Hospital, Incheon
  - Park Urology Clinic, Incheon
  - Hanvit Urology Clinic, Incheon
  - Lee and Lee dermatology urology clinic, Incheon
  - Songdo Hospital, Seoul
  - Dr. Cho & Lee's Urology Clinic, Seoul
  - Won Urology Clinic, Seoul
  - Lim Urology Clinic, Seoul
  - Dong Seoul Hospital, Seoul
  - Woo Tae Hyung urology clinic, Seoul
  - S-Up Clinic, Seoul
  - Park Yong Hyun Urology Clinic, Seoul
  - Saerom urology clinic, Seoul
  - Park Kyu Hong Urology Clinic, Seoul
  - Seonreung Top Urology Clinic, Seoul
  - Yonsei Woono Urology Clinic, Seoul
  - Daehang Hospital, Seoul
  - Park Byung Dae Urology Clinic, Seoul
  - Jin Kilnam Urology Clinic, Seoul
  - Bes Top Urology Clinic, Seoul
  - Song Woung Soeg Urology Clinic, Seoul
  - Kim Jun-Ho Urology Clinic, Seoul
  - Hong Don Ho Urology Clinic, Seoul
  - Boram St.Mary's Internal Medicine, Seoul
  - Nowon Paik Urology Clinic, Seoul
  - Su clinic, Seoul
  - Uh's Urology Clinic, Seoul
  - Seoul Top Clinic, Seoul
  - Urotop Urology Clinic, Seoul
  - Yoo Jong Keun Urology Clinic, Seoul
  - Seong Ae Hospital, Seoul
  - Korea Ace Urology Clinic, Seoul
  - Woo ri dermatology urology clinic, Seoul
  - Bae Urology Hospital, Seoul
  - Jung Ho Hyun Urology Clinic, Seoul
  - Miz-Medi Hospital, Seoul
  - Choi Urology Hospital, Seoul
  - Ulsan Jeil Hopital, Ulsan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0221075&StudyName=Toviaz%20Post%20Marketing%20Surveillance%20Study

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between November 2009 and August 2014 from 235 Korean medical care centers.
Groups:
- Toviaz: Participants were administered with Toviaz as part of routine care. The use and dosage recommendations for Toviaz were based on the approved local product document and were adjusted solely according to medical and therapeutic necessity.
Period: Overall Study
Arm/Group | Toviaz
Started | 3109
Completed | 2434
Not Completed | 675
Not completed — Visit Stop | 399
Not completed — Lack of Efficacy | 64
Not completed — Adverse Event | 41
Not completed — Other Reasons | 171

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: regardless of treatment period, all participants who received study drug once or more, including dropouts due to adverse event (AE), were included in the safety analysis set. Participants who started Toviaz prior to the contract date or violated usage of maximum daily dose of 8 mg were excluded from the safety analysis set.
Arm/Group | Toviaz
Number analyzed (Participants) | 3107
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.22 (13.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1520
  Male | 1587

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence in a clinical investigation subject administered a product or medical device; the event was not necessarily had a causal relationship with the treatment or usage. All AEs reported after start of administration of Toviaz were considered as TEAEs.
Time Frame: From the time that the participant signed data privacy statement through and including 28 calendar days after the last administration of the study drug.
Population: Safety Analysis Set
Measure: Number; unit: Percentage of Participants
Arm/Group | Toviaz
Number analyzed (Participants) | 3107
Percentage of Participants | 8.53

2. Primary Outcome: Investigator's Final Assessment of Effectiveness at the End of Study Treatment
Description: The final efficacy assessment included improvement, no change, aggravation, and unevaluable evaluated by the investigator based on the subject's symptoms of frequent micturition, urgency, and urgency urinary incontinence (UUI).
Time Frame: At the end of study treatment
Population: Per-Protocol (PP) Population: participants who had evaluable data and were eligible for the efficacy assessment of the approved indication. The method of last observation carried forward was used in the analysis of effectiveness endpoints.
Measure: Number; unit: Percentage of Participants
Arm/Group | Toviaz
Number analyzed (Participants) | 2978
Percentage of Participants
  Improvement | 90.13
  No Change | 9.50
  Aggravation | 0.37

3. Secondary Outcome: Change From Baseline in Number of Micturitions Per 24 Hours at the End of Study Treatment
Description: The number of micturitions per 24 hours was recorded in the case report form (CRF) by the investigator. Baseline was defined as data collected within 1 week prior to the first visit.
Time Frame: Baseline and at the end of study treatment
Population: PP Population; n refers to the number of participants with evaluable data.
Measure: Mean (Standard Deviation); unit: Number of Episodes per 24 Hours
Arm/Group | Toviaz
Number analyzed (Participants) | 2718
Number of Episodes per 24 Hours
  Baseline (n=2718) | 12.05 (3.20)
  End of Study Treatment (n=2718) | 8.04 (2.35)
  Change from Baseline (n=2718) | -4.02 (2.66)
Statistical Analysis 1: Comparison: Toviaz; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Statistical significant level: 0.05

4. Secondary Outcome: Change From Baseline in Number of Urgency Episodes Per 24 Hours at the End of Study Treatment
Description: The number of urgency episodes per 24 hours was recorded in the CRF by the investigator. Baseline was defined as data collected within 1 week prior to the first visit.
Time Frame: Baseline and at the end of study treatment
Population: PP Population; n refers to the number of participants with evaluable data.
Measure: Mean (Standard Deviation); unit: Number of Episodes per 24 Hours
Arm/Group | Toviaz
Number analyzed (Participants) | 2724
Number of Episodes per 24 Hours
  Baseline (n=2724) | 3.65 (3.58)
  End of Study Treatment (n=2724) | 1.27 (2.05)
  Change from Baseline (n=2724) | -2.37 (2.67)
Statistical Analysis 1: Comparison: Toviaz; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Statistical significant level: 0.05

5. Secondary Outcome: Change From Baseline in Number of UUI Episodes Per 24 Hours at the End of Study Treatment
Description: The number of UUI episodes per 24 hours was recorded in the CRF by the investigator. Baseline was defined as data collected within 1 week prior to the first visit.
Time Frame: Baseline and at the end of study treatment
Population: PP Population; n refers to the number of participants with evaluable data.
Measure: Mean (Standard Deviation); unit: Number of Episodes per 24 Hours
Arm/Group | Toviaz
Number analyzed (Participants) | 2800
Number of Episodes per 24 Hours
  Baseline (n=2800) | 1.07 (2.05)
  End of study treatment (n=2800) | 0.27 (0.89)
  Change from baseline (n=2800) | -0.80 (1.65)
Statistical Analysis 1: Comparison: Toviaz; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Statistical significant level: 0.05

6. Secondary Outcome: Participant Perception of Bladder Condition at the End of Study Treatment
Description: Participant perception of bladder condition was recorded in the CRF by the investigator. Participants were asked at baseline (BL) and at the end of study treatment (EOT) if the extent to which their bladder condition caused them problems. The possible responses were: No Problem, Very Minor Problems, Minor Problems, Moderate Problems, Severe Problems, or Many Severe Problems.
Time Frame: Baseline and at the end of study treatment
Population: PP Population
Measure: Number; unit: Participants
Arm/Group | Toviaz
Number analyzed (Participants) | 2939
Participants
  BL: No Problem/EOT: No problem | 0
  BL: No Problem/EOT: Very Minor Problems | 0
  BL: No Problem/EOT: Minor Problems | 0
  BL: No Problem/EOT: Moderate Problems | 1
  BL: No Problem/EOT: Severe Problems | 0
  BL: No Problem/EOT: Many Severe Problems | 0
  BL: Very Minor Problems/EOT:No Problem | 29
  BL:Very Minor Problems/EOT: Very Minor Problems | 33
  BL: Very Minor Problems/EOT: Minor Problems | 0
  BL: Very Minor Problems/EOT: Moderate Problems | 0
  BL: Very Minor Problems/EOT: Severe Problems | 0
  BL: Very Minor Problems/EOT: Many Severe Problems | 0
  BL: Minor Problems/EOT: No Problem | 105
  BL: Minor Problems/EOT: Very Minor Problems | 134
  BL: Minor Problems/EOT: Minor Problems | 42
  BL: Minor Problems/EOT:Moderate Problems | 1
  BL: Minor Problems/EOT: Severe Problems | 0
  BL: Minor Problems/EOT: Many Severe Problems | 0
  BL: Moderate Problems/EOT: No Problem | 224
  BL: Moderate Problems/EOT: Very Minor Problems | 447
  BL: Moderate Problems/EOT: Minor Problems | 171
  BL: Moderate Problems/EOT: Moderate Problems | 116
  BL: Moderate Problems/EOT: Severe Problems | 3
  BL: Moderate Problems/EOT: Many Severe Problems | 1
  BL: Severe Problems/EOT: No Problem | 188
  BL: Severe Problems/EOT: Very Minor Problems | 456
  BL: Severe Problems/EOT: Minor Problems | 227
  BL: Severe Problems/EOT: Moderate Problems | 97
  BL: Severe Problems/EOT: Severe Problems | 49
  BL: Severe Problems/EOT: Many Severe Problems | 0
  BL: Many Severe Problems/EOT: No Problem | 105
  BL: Many Severe Problems/EOT: Very Minor Problems | 195
  BL: Many Severe Problems/EOT: Minor Problems | 148
  BL: Many Severe Problems/EOT: Moderate Problems | 97
  BL: Many Severe Problems/EOT: Severe Problems | 51
  BL: Many Severe Problems/EOT: Many Severe Problems | 19

7. Secondary Outcome: Percentage of Participants With a Final Efficacy Assessment of Effective by Baseline and Treatment Characteristics
Description: Participants who were assessed as having improved from their baseline condition in the final efficacy assessment were considered as "effective". Baseline and treatment characteristics included: geriatric status (<65 years or ≥65 years), age categories, gender, weight categories, height categories, allergic history, duration of disease, past overactive bladder (OAB) treatment history, medical history, kidney and liver disorders, concomitant medication, total administration period of Toviaz, completion status, daily dose of Toviaz, and long term administration of Toviaz (<274 days and ≥274 days) .
Time Frame: At the end of study treatment
Population: PP Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Toviaz
Number analyzed (Participants) | 2978
Percentage of Participants
  All Participants | 90.13 [89.06 to 90.15]
  Geriatric Status: <65 years | 90.86 [89.47 to 90.89]
  Geriatric Status: ≥65 years | 89.20 [87.52 to 89.25]
  Age Category: <50 years | 91.27 [89.07 to 91.36]
  Age Category: 50 to 59 years | 91.08 [88.87 to 91.17]
  Age Category: 60 to 69 years | 89.29 [87.22 to 89.36]
  Age Category: 70 to 79 years | 89.45 [87.13 to 89.54]
  Age Category: ≥80 years | 89.27 [84.71 to 89.61]
  Gender: Male | 88.98 [87.41 to 89.02]
  Gender: Female | 91.36 [89.91 to 91.40]
  Weight Category: <50 kg | 89.73 [85.36 to 90.05]
  Weight Category: 50 to <60 kg | 91.64 [89.72 to 91.70]
  Weight Category: 60 to <70 kg | 90.32 [88.47 to 90.38]
  Weight Category: ≥70 kg | 88.82 [86.59 to 88.90]
  Height Category: <160 cm | 89.99 [87.93 to 90.06]
  Height Category: 160 to 170 cm | 90.32 [88.57 to 90.37]
  Height Category: ≥170 cm | 90.35 [88.33 to 90.42]
  Allergic History: Yes | 82.22 [71.05 to 83.89]
  Allergic History: No | 90.25 [89.18 to 90.27]
  Duration of Disease: <1 week | 92.40 [91.18 to 92.43]
  Duration of Disease: 1 to <8 weeks | 89.42 [85.90 to 89.63]
  Duration of Disease: 8 to <16 weeks | 89.05 [83.82 to 89.50]
  Duration of Disease: ≥16 weeks | 84.33 [81.54 to 84.44]
  Past OAB Treatment History: Yes | 85.30 [82.79 to 85.39]
  Past OAB Treatment History: No | 91.79 [90.64 to 91.81]
  Existence for Medical History of Past Disease: Yes | 87.96 [84.80 to 88.12]
  Existence for Medical History of Past Disease: No | 90.47 [89.34 to 90.49]
  Medical History of Present Disease: Yes | 87.96 [86.34 to 88.00]
  Medical History of Present Disease: No | 92.46 [91.10 to 92.50]
  Kidney Disease: Yes | 90.00 [71.41 to 95.88]
  Kidney Disease: No | 90.13 [89.05 to 90.15]
  Liver Disorder: Yes | 92.31 [77.82 to 96.33]
  Liver Disorder: No | 90.12 [89.04 to 90.14]
  Administration Period of Toviaz: <2 months | 85.22 [82.96 to 85.29]
  Administration Period of Toviaz: 2 to <4 months | 92.44 [91.16 to 92.47]
  Administration Period Of Toviaz: ≥ 4 months | 92.33 [89.64 to 92.47]
  Daily Dose of Toviaz: 3 mg | 66.67 [13.32 to 97.47]
  Daily Dose of Toviaz: 4 mg | 90.65 [89.51 to 90.68]
  Daily Dose of Toviaz: >4 to <8 mg | 85.25 [80.80 to 85.53]
  Daily Dose of Toviaz: 8 mg | 90.25 [86.47 to 90.50]
  Completion | 92.28 [91.22 to 92.30]
  Discontinuation | 80.72 [77.44 to 80.86]
  Total Administration Period <274 days | 90.16 [89.09 to 90.18]
  Total Administration Period ≥274 days | 87.50 [77.25 to 89.12]
  Existence for Concurrent Medication: Yes | 88.48 [86.92 to 88.51]
  Existence for Concurrent Medication: No | 92.08 [90.65 to 92.12]
Statistical Analysis 1: Comparison: Toviaz; Geriatric Status: <65 years versus (vs) Geriatric Status: ≥65 years; Test type: Superiority or Other; p = 0.1319, Chi-squared — Statistical significant level: 0.05
Statistical Analysis 2: Comparison: Toviaz; Comparison among Age Categories: <50 years, 50 to 59 years, 60 to 69 years, 70 to 79 years, and ≥80 years; Test type: Superiority or Other; p = 0.6010, Chi-squared — Statistical significant level: 0.05
Statistical Analysis 3: Comparison: Toviaz; Male vs Female; Test type: Superiority or Other; p = 0.0289, Chi-squared — Statistical significant level: 0.05
Statistical Analysis 4: Comparison: Toviaz; Comparison among Weight Categories: <50 kg, 50 to 60 kg, 60 to 70 kg, and ≥70 kg; Test type: Superiority or Other; p = 0.3078, Chi-squared — Statistical significant level: 0.05
Statistical Analysis 5: Comparison: Toviaz; Comparison among Height Categories: <160 cm, 160 to 170 cm, and ≥170 cm; Test type: Superiority or Other; p = 0.9614, Chi-squared — Statistical significant level: 0.05
Statistical Analysis 6: Comparison: Toviaz; Allergic History: Yes vs Allergic History: No; Test type: Superiority or Other; p = 0.0788, Fisher Exact — Statistical significant level: 0.05
Statistical Analysis 7: Comparison: Toviaz; Comparison among Duration of Disease: <1 week, 1 to 8 weeks, 8 to 16 weeks, and ≥16 weeks; Test type: Superiority or Other; p < 0.0001, Chi-squared — Statistical significant level: 0.05
Statistical Analysis 8: Comparison: Toviaz; Past OAB Treatment History: Yes vs Past OAB Treatment History: No; Test type: Superiority or Other; p < 0.0001, Chi-squared — Statistical significant level: 0.05
Statistical Analysis 9: Comparison: Toviaz; Medical History of Past Disease: Yes vs Medical History of Past Disease: No; Test type: Superiority or Other; p = 0.1147, Chi-squared — Statistical significant level: 0.05
Statistical Analysis 10: Comparison: Toviaz; Medical History of Present Disease: Yes vs Medical History of Present Disease: No; Test type: Superiority or Other; p < 0.0001, Chi-squared — Statistical significant level: 0.05
Statistical Analysis 11: Comparison: Toviaz; Kidney Disorder: Yes vs Kidney Disorder: No; Test type: Superiority or Other; p = 1.0000, Fisher Exact — Statistical significant level: 0.05
Statistical Analysis 12: Comparison: Toviaz; Liver Disorder: Yes vs Liver Disorder: No; Test type: Superiority or Other; p = 1.0000, Fisher Exact — Statistical significant level: 0.05
Statistical Analysis 13: Comparison: Toviaz; Comparison among Total Administration Period of Toviaz Subgroups: <2 months, 2 to 4 months, and ≥4 months; Test type: Superiority or Other; p < 0.0001, Chi-squared — Statistical significant level: 0.05
Statistical Analysis 14: Comparison: Toviaz; Comparison among Daily Dose of Toviaz: 3 mg, 4 mg, >4 mg to <8 mg, and 8 mg; Test type: Superiority or Other; p = 0.0239, Fisher Exact — Statistical significant level: 0.05
Statistical Analysis 15: Comparison: Toviaz; Completion vs Discontinuation; Test type: Superiority or Other; p < 0.0001, Chi-squared — Statistical significant level: 0.05
Statistical Analysis 16: Comparison: Toviaz; Total Administration Period <274 days vs Total Administration Period ≥ 274 days; Test type: Superiority or Other; p = 0.5889, Fisher Exact — Statistical significant level: 0.05
Statistical Analysis 17: Comparison: Toviaz; Concurrent Medication: Yes vs Concurrent Medication: No; Test type: Superiority or Other; p = 0.0010, Chi-squared — Statistical significant level: 0.05

ADVERSE EVENTS:
Time Frame: From the time that the participant signed data privacy statement through and including 28 calendar days after the last administration of the study drug.
Description: The same event may appear as both an AE and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another participant, or 1 participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Toviaz
Serious Adverse Events (participants affected / at risk) | 0/3107
Other Adverse Events (participants affected / at risk) | 219/3107
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Toviaz (N=3107)
Constipation (Gastrointestinal disorders) | 48
Mouth dry (Gastrointestinal disorders) | 168
Micturition disorder (Renal and urinary disorders) | 35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days